CLINICAL TRIAL: NCT06310382
Title: A Phase I/II Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Antitumor Activity of GH55 in Patients Harboring MAPK Pathway Mutations in Advanced Solid Tumors
Brief Title: GH55 for Advanced Cancers With MAPK Mutations: A Study on Safety and Early Results
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Genhouse Bio Co., Ltd. (Other)
Collaborators: Shanghai East Hospital (Other); Shandong Tumor Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GH55-CRS001
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Tumors With MAPK Signal Pathway Mutations

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GH55 GROUP (Experimental)
  Interventions: Drug: GH55

INTERVENTIONS:
Drug: GH55 — GH55 capsule is a novel small molecule, highly selective dual-mechanism ERK1/2 inhibitor developed by Suzhou Genhouse Bio. Co., Ltd. This product can be used to treat cancers caused by abnormal activation of the MAPK pathway (mutational activation of RAS/RAF/MEK) by targeted inhibition of ERK1/2.

SUMMARY:
This is a multi-center, open-label, dose escalation phase I and dose expansion phase II study aimed to evaluate the safety, tolerability, PK and PD profiles as well as to observe the efficacy of GH55 in patients with MAPK mutant advanced solid tumors.

This study is divided into two parts, namely the dose escalation phase I study and the dose expansion phase II study.

DETAILED DESCRIPTION:
This study is divided into two parts, namely the dose escalation phase I study and the dose expansion phase II study. This study plans to include 5 dose groups, namely 40 mg, 80 mg, 150 mg, 200 mg, and 250 mg, and adopts a "3+3" dose escalation design. All of the 40 mg, 80 mg, 150 mg, 200 mg and 250 mg groups will adopt the "3+3" design, and 3-6 subjects will be enrolled in each group. The enrollment of the first subject and subsequent subject in each dose group should be at least 7 days apart.

Subjects will receive a single dose of GH55 on day 1 (Cycle 0 Day 1, C0D1). The investigator will assess the safety data on day 3 (C0D3) to determine whether subjects can be initiated on multiple doses of GH55 [quaque die (QD) continuously, and 3 weeks per cycle] on day 4 (C1D1). The dose limiting toxicity (DLT) observation period is from the initiation of single dosing to the end of the first cycle of multiple dosing [Cycle 0 (3 days) and Cycle 1 (3 weeks)]. The sponsor and investigator will jointly assess the safety data to determine whether to ascend to the next higher dose. These steps will be repeated until MTD is reached, and the safety, tolerability, and PK profile of single dose and multiple doses of oral administration of GH55 will be assessed. If MTD cannot be determined when the dose escalation study is complete, the sponsor and investigator will jointly determine whether to increase the ascending dose based on the existing safety, tolerability, PK, PD and preliminary efficacy data. All subjects can continue the treatment until disease progression, initiation of new antitumor treatment, withdrawal of informed consent, or death (whichever occurs first). The dose expansion phase II study will begin once the last subject in the dose escalation phase I study has completed the DLT observation. Two dose expansion groups will be designed, with a dose level in each group that is expected to become the RP2D based on the safety, tolerability, PK/PD profile, and preliminary efficacy data of GH55 in the dose escalation phase I study. Two dose expansion groups will enroll 60-80 subjects to further evaluate the efficacy, safety, and PK/PD profile of GH55 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following inclusion criteria to be qualified for study enrollment:

1. Male or female subjects aged 18-80 years (inclusive).
2. Patients with histologically or cytologically confirmed MAPK mutant (presence of RAS/RAF/MEK/ERK mutations) locally advanced or metastatic solid tumors.
3. Patients who have failed standard treatment or have no standard treatment regimen or are not suitable for standard treatment currently.
4. Dose escalation: At least one assessable tumor lesion according to RECIST version 1.1; Dose expansion: At least one measurable tumor lesion according to RECIST version 1.1 (tumor lesion located in the region of previous radiotherapy or other locoregional treatment sites is usually not considered a measurable lesion, unless this lesion shows clear progression or persists for 3 months after radiotherapy).
5. Eastern Cooperative Oncology Group (ECOG) performance status score: Phase I dose escalation: 0-1. Phase II dose expansion: 0-2.
6. 3 months or longer expected survival.
7. Major organs are functioning normally, and laboratory tests meet the following criteria during the screening period.

Hematological system (has not received any blood transfusion or hematopoietic stimulating factor therapy within the past 14 days) Absolute neutrophil count (ANC) ≥ 1.5 × 109/L Platelet Count (PLT) ≥ 75 × 109/L Hemoglobin (Hb) ≥ 90 g/L Liver function Albumin (ALB) ≥ 3.0 g/dL Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN) Liver metastasis or liver cancer patients: ≤ 2.5 × ULN Alanine Aminotransferase (ALT) ≤ 2.5 × ULN; Liver metastasis or liver cancer patients: ≤ 5 × ULN Aspartate aminotransferase (AST) ≤ 2.5 × ULN; Liver metastasis or liver cancer patients: ≤ 5 × ULN Renal function Creatinine clearance rate (Ccr) ≥ 60 mL/min (calculated based on the Cockcroft-Gault formula) Coagulation function Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN International normalized ratio (INR) ≤ 1.5 × ULN Cardiac function Left ventricular ejection fraction (LVEF) ≥ 50% QT interval corrected by the Fridericia formula (QTcF) Males < 450 ms, Females < 470 ms 7. Qualified patients (male and female) with childbearing potential must agree to use reliable contraceptives (hormone or barrier or abstinence) with their partners during the study and until at least 3 months after the last dose; female patients with childbearing potential must be negative for the blood pregnancy test within 1 week before the first dose.

8. Subjects must give informed consent to the study and voluntarily signed the informed consent form prior to study initiation.

Exclusion Criteria:

Subjects who meet any one of the following exclusion criteria are not eligible for study enrollment:

1. Received antitumor therapy such as chemotherapy within 3 weeks before the first dose, radiotherapy, biotherapy, endocrine therapy, targeted therapy, and immunotherapy within 4 weeks before the first dose, except for the following:

   * Use of nitrosoureas or mitomycin C within 6 weeks prior to the first dose of the investigational drug;
   * Use of oral fluorouracil(s), small molecule targeted drugs, and antitumor traditional Chinese medicine within 2 weeks prior to the first dose of the investigational drug;
   * Local palliative radiotherapy within 2 weeks prior to the first dose of the investigational drug.
2. Received other unmarketed clinical investigational drug or therapy within 4 weeks prior to the first dose.
3. Underwent major organ surgery (excluding needle biopsy) or had significant trauma within 4 weeks prior to the first dose or requires selective surgery during the study period.
4. Use of strong CYP3A4 inhibitors or inducers within 1 week prior to the first dose of the investigational drug.
5. Previously received other selective ERK inhibitors.
6. Previously received allogeneic HSCT or organ transplantation.
7. Adverse drug reactions of previous antitumor treatment have not recovered to grade ≤ 1 as per CTCAE version 5.0 (except for toxicity without safety risk judged by the investigator, such as alopecia, grade 2 peripheral neurotoxicity, and hypothyroidism that is stable after hormone replacement therapy).
8. Brain parenchymal metastasis or meningeal metastasis with clinical symptoms unsuitable for study participation as judged by the investigator.
9. Patient with active infection and currently requires intravenous anti-infective therapy.
10. History of immunodeficiency, including being positive for HIV antibody test.
11. Active hepatitis B [HBsAg positive and HBV-DNA > 500 IU/mL or LLQ of the study site (when the LLQ is > 500 IU/mL)], for which antiviral therapies other than interferon are permitted; Active hepatitis C (patients who are positive for HCV antibody but whose HCV-RNA is < study site LLQ can be included).
12. History of severe cardiovascular and cerebrovascular diseases, including but not limited to:

    * Severe abnormalities in cardiac rhythm or conduction, such as ventricular arrhythmia or second- or third-degree atrioventricular block requiring clinical intervention;
    * Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other grade 3 or greater cardiovascular and cerebrovascular events within 6 months prior to the first dose;
    * New York Heart Disease Association (NYHA) class ≥ III cardiac function or left ventricular ejection fraction (LVEF) < 50%;
    * Clinically uncontrolled hypertension;
    * Any factors that increase the risk of QTc prolongation or arrhythmia, such as heart failure, hypokalemia that is difficult to correct, congenital long QT syndrome, family history of long QT syndrome, and use of concomitant medication known to prolong QT interval.
13. History of other malignant tumors (except for the cured squamous cell carcinoma in situ of the skin, basal cell carcinoma, and cervical carcinoma in situ that have not recurred within 5 years and are considered acceptable for study enrollment by the investigator; except for patients who are considered acceptable for enrollment by the investigator in the dose escalation study).
14. History of retinal vein occlusion or central serous retinopathy, or patients with clinically significant abnormalities in the ophthalmological examination during the screening period and judged by the investigator to be unsuitable for enrollment.
15. Unable to swallow medication or has conditions that severely impact gastrointestinal absorption (e.g. Chronic diarrhea or intestinal obstruction) as judged by the investigator.
16. Clinically uncontrolled third space effusion judged by the investigator to be unsuitable for enrollment.
17. Patients with current interstitial lung disease (except radiation-induced pulmonary fibrosis that does not required hormone therapy).
18. Known alcohol or drug dependence.
19. Mental disorder or poor compliance.
20. Previous history of severe allergy, or allergy to any active or non-active ingredients of the investigational drug.
21. Pregnant or lactating women.
22. Other conditions judged by the investigator that render the subject unsuitable for participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2025-05-26 (Estimated); Study Completion 2025-08-04 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicities Incidence Count Among Study Participants | 2 years
  Incidence of dose limiting toxicities (DLTs) in the dose escalation phase. A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first treatment cycle. (phase I)
Number of Participants Reporting Adverse Events (AEs) or Serious Adverse Events (SAEs)Objective | 2 years
  All patients participating in this study will be assessed for incidence and severity of adverse events (AEs) and serious AEs, including changes in laboratory values, vital signs, electrocardiograms, cardiac imaging and ophthalmological assessments (phase I)
Response Rate (ORR) Based on RECIST 1.1 Criteria | 2 years
  ORR is defined as the proportion of participants with complete response or partial response (CR+PR). (phase II)

SECONDARY OUTCOMES:
Progression-free survival (PFS) Based on RECIST 1.1 Criteria | 2 years
  PFS is defined as the interval of time between the date of first treatment to the earliest date of disease progression or death which occurs first. (phase I/II)
Duration of response (DOR) Based on RECIST 1.1 Criteria | 2 years
  DCR is defined as proportion of participants with complete response, partial response, stable disease(CR+PR+SD). (phase I/II)
Number of participants with adverse events | 2 years
  All patients participating in this study will be assessed for incidence and severity of adverse events (AEs) and serious AEs, including changes in laboratory values, vital signs, electrocardiograms, cardiac imaging and ophthalmological assessments (phase II)
Plasma concentration (Cmax) | 2 years
  Highest observed plasma concentration of GH55. (phase I/II)
Time to achieve Cmax (Tmax) | 2 years
  Time of highest observed plasma concentration of GH55. (phase I/II)
Area under the plasma concentration-time curve (AUC) | 2 years
  Area under the plasma concentration time curve of GH55. (phase I/II)

CONTACTS AND LOCATIONS:
Overall Officials: JIN LI, DPCTORATE, Principal Investigator — 021-38804518; HAIDAN WANG, DOCTORATE, Study Director — 0512-86861608
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China